CLINICAL TRIAL: NCT03275649
Title: Development of an Intervention to Increase Help-seeking for Non-motor Symptoms in People With Parkinson's
Brief Title: Help-seeking for Health Problems in People With Parkinson's
Acronym: PDHelp
Status: Completed | Type: Observational
Sponsor: City, University of London (Other)
Collaborators: King's College London (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CityULondon_PDHelp
Record Dates: First submitted 2017-08-29; First posted 2017-09-07 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Help-seeking for non-motor symptoms — Brief, self-paced, online individually tailored intervention using LifeGuide software. Includes information, videos and exercises.

SUMMARY:
Non-motor symptoms (NMS) are common in Parkinson's disease (PD) and cause significant distress and decreased quality of life. A high rate of non-declaration of NMS by patients means that many NMS remain unrecognized and untreated, even in specialist clinical services. In phase one of this research qualitative interviews (phase 1) were guided by the Theoretical Domains Framework and used to identify the barriers for help-seeking. A quantitative questionnaire survey (phase 2) examined the significance of these barriers to help seeking. The present study aims to develop (phase 3) and test the feasibility (phase 4) of a targeted behavioural intervention of barriers which were identified in phases 1 and 2 which prevent help-seeking for NMS in patients with PD. As with phases 1 and 2, the feasibility trial will include people with unreported burdensome NMS, who have not reported them to their PD consultant or nurse. The intervention has been co-designed by people affected by Parkinson's and targets the barriers identified in the previous phases of the research. In phase three of the research, 'think-aloud' interviews will be used to further develop the intervention so that it is acceptable and easy to use. In the final phase, a feasibility trial will be conducted to examine efficacy of the intervention for increasing help-seeking for undeclared NMS. The study has implications for using a theoretically driven behavioural intervention to promote help-seeking for NMS and ultimately increase receipt of clinical care for NMS among patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's
* Access to a computer and internet connection
* Experiencing at least one unreported non-motor symptom

Exclusion Criteria:

* Presence of sensory loss or communication difficulty (including inadequate command of English) sufficient to interfere with the assessments.
* Severe cognitive impairment that would make participation in the intervention problematic or distressing. This will be assessed using the Telephone Interview for Cognitive Status-Modified (TICS-M, Brandt et al., 1993). People with a score of less than 20 will be excluded.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: -Participants diagnosed with idiopathic PD will be recruited through outpatient neurology clinics and via the Parkinson's UK research network. Participants experiencing burdensome undisclosed non-motor symptoms will be recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients help-seeking post-intervention | 1 week
  after intervention

SECONDARY OUTCOMES:
Number of eligible patients completing the study | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- City, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided